CLINICAL TRIAL: NCT06225895
Title: Bilateral Rhomboid Intercostal Block Versus Erector Spinae Plane Block for Perioperative Analgesia in Patients Undergoing Bilateral Reduction Mammoplasty
Brief Title: Bilateral Rhomboid Intercostal Block for Perioperative Analgesia in Patients Undergoing Bilateral Reduction Mammoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, associate professor of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11408//15-1-2024
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Analgesia
Keywords: Rhomboid Intercostal Block; Erector Spinae Plane Block; Reduction Mammoplasty; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, General; Bupivacaine

STUDY DESIGN:
Intervention Model Description: computer generating random numbers, the patients will be allocated into three equal groups: Group C: (control group) patients will receive general anesthesia. Group E: patients will receive an Erector spinea plane block with 20 ml of bupivacaine 0.25% on each side followed by general anesthesia.
  Group R: patients will receive rhomboid intercostal nerve block with 20 ml of bupivacaine 0.25% on each side followed by general anesthesia.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) double-blinded(participants and outcome assessors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Placebo Comparator): patients will receive general anesthesia
  Interventions: Procedure: general anesthesia
- E group (Active Comparator): patients will receive Erector spinae plane block
  Interventions: Procedure: general anesthesia; Procedure: Erector spinae plane block; Drug: Bupivacaine
- R group (Active Comparator): patients will receive rhomboid intercostal nerve block
  Interventions: Procedure: general anesthesia; Procedure: a rhomboid intercostal nerve block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: general anesthesia — patients will receive general anesthesia.
Procedure: Erector spinae plane block — patients will receive Erector spinae plane block with 20 ml of bupivacaine 0.25% on each side followed by general anesthesia.
  Arms: E group
Procedure: a rhomboid intercostal nerve block — patients will receive a rhomboid intercostal nerve block with 20 ml of bupivacaine 0.25% on each side followed by general anesthesia.
  Arms: R group
Drug: Bupivacaine — 20 ml of bupivacaine 0.25%
  Arms: E group; R group

SUMMARY:
Bilateral reduction mammoplasty is one of the most commonly performed breast surgery. The Postoperative pain following it should be minimized.

Opioid administration for acute pain after reduction mammoplasty surgery has many side effects. Regional block techniques such as paravertebral block and thoracic epidural anesthesia have possible complications and technical difficulties.

The new alternative regional techniques such as erector spinae plane block and rhomboid intercostal plane block are clinical trials for providing a safe, easy, and painless anesthetic procedure with adequate postoperative analgesia for a large section of patients undergoing thoracic surgeries.

DETAILED DESCRIPTION:
Reduction mammoplasty is the gold standard procedure for symptomatic breast hypertrophy and it is also used for contralateral breast symmetrisation following breast cancer surgery. Symptomatic hypermastia affects the quality of life of millions of women worldwide. The most frequent symptoms shown by more than two-thirds of patients are shoulder grooving, and back, shoulder, and neck pain. Reduction mammoplasty proved to be an effective treatment, both aesthetically and functionally, with a demonstrated consistently high patient satisfaction.

Optimal pain management is an essential component of enhanced recovery after surgery protocols that are becoming standard of care because they have been shown to reduce postoperative complications and expedite recovery. However, postoperative pain is still inadequately managed. Opioids remain the mainstay of perioperative pain management, despite well-recognized adverse events including nausea, vomiting, pruritus, and respiratory depression.

Regional anesthesia has been believed as one of the formats for effective perioperative pain control. Plane blocks such as the serratus anterior plane (SAP) block, pectoral nerve block, and erector spinae plane block have gained popularity during multimodal analgesia after various surgical procedures.

The erector spinae plane block (ESPB) was initially introduced by Forero et al. in 2016 and offers extensive analgesia in thoracic surgery. It can be used as a substitute for PVB because it is less intrusive, simpler, and safer to apply plane blocks that are applied in the plane of the spine's erector muscles.

Rhomboid intercostal block (RIB) was described in 2016 as an alternative to thoracic epidural analgesia. The local anesthetic agent is delivered into the plane between the rhomboid major and intercostal muscles. That provides good analgesia for the anterior and posterior hemithorax.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Age 18-65 years old.
* BMI ≤ 35 kg/m2
* ASA I - II.
* Elective bilateral reduction mammoplasty surgery under general anesthesia.
* Duration of surgery within five hours

Exclusion Criteria:

* Patients on anti-platelet, anticoagulant, or B blocker drugs.
* Patients with acute decompensated heart failure, hypertension, heart block, coronary disease, Asthma
* History of allergy to the local anesthetics (LA) agents used in this study,
* Skin lesion at the needle insertion site,
* Those with bleeding disorders, sepsis, liver disease, psychiatric disorders, and pregnancy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This surgery is only performed for women
Enrollment: 72 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Time to first dose of rescue analgesia | in the first postoperative 24 hours
  is the time from the end of operation to patient reporting VAS ≥ 3. Thereafter, rescue analgesia in the form of 0.1mg/kg IV of nalbuphine will be injected.
Total nalbuphine consumption | in the first 24 hours postoperatively
  total dose of nalbuphine rescue analgesic that the patient required postoperatively

SECONDARY OUTCOMES:
changes of pain assessment | at 1hour, 3,6,12, 24 hours postoperatively
  visual analogue scale will be recorded at rest and movement
non invasive blood pressure | immediately prior to surgery, immediately after skin incision, 15,30,60,120,180,240 min intraoperatively and at end of surgery
  changes of hemodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Shereen E Abd Ellatif, M.D., Principal Investigator — Faculty of medicine, zagazig university
Locations (2):
- Egypt (2):
  - Faculty of medicine, zagazig university, Zagazig, Alsharqia
  - Shereen E Abd Ellatif, Zagazig, Alsharqia

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: planned after the completion of the study and publication
Access Criteria: contact with principal investigatoR

REFERENCES:
- [Background] Gad M, Abdelwahab K, Abdallah A, Abdelkhalek M, Abdelaziz M. Ultrasound-Guided Erector Spinae Plane Block Compared to Modified Pectoral Plane Block for Modified Radical Mastectomy Operations. Anesth Essays Res. 2019 Apr-Jun;13(2):334-339. doi: 10.4103/aer.AER_77_19. PMID 31198256
- [Background] Viscardi JA, Oranges CM, Schaefer DJ, Kalbermatten DF. Reduction Mammoplasty: A Ten-Year Retrospective Review of the Omega Resection Pattern Technique. J Clin Med. 2021 Sep 27;10(19):4418. doi: 10.3390/jcm10194418. PMID 34640438
- [Background] Elsharkawy H, Saifullah T, Kolli S, Drake R. Rhomboid intercostal block. Anaesthesia. 2016 Jul;71(7):856-7. doi: 10.1111/anae.13498. No abstract available. PMID 27291611
- [Background] Tunay DL, Ilginel MT, Karacaer F, Biricik E, Tabakan I, Ozmete O. Bilateral Ultrasound-Guided Erector Spinae Plane Block for Perioperative Analgesia in Breast Reduction Surgery: A Prospective Randomized and Controlled Trial. Aesthetic Plast Surg. 2023 Aug;47(4):1279-1288. doi: 10.1007/s00266-023-03315-0. Epub 2023 Mar 16. PMID 36928313
- [Background] Yayik AM, Ahiskalioglu A, Ates I, Ahiskalioglu EO, Cinal H. Ultrasound guided bilateral rhomboid intercostal block for breast reduction surgery. J Clin Anesth. 2019 Nov;57:38-39. doi: 10.1016/j.jclinane.2019.03.001. Epub 2019 Mar 6. No abstract available. PMID 30851503